CLINICAL TRIAL: NCT04177329
Title: Impact of Cardiac Complications on Outcomes of Patients After Subarachnoid Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reda Omar, princible investegator Resident doctor at neuro_psychiatry department, Assiut University
Other Study IDs: Impact of cardiac complication
Record Dates: First submitted 2019-09-23; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with subarachnoid haemorrhage frequently develop cardiac complications affecting their outcome

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as spontaneous subarachnoid hemorrhage.
* SSAH patients aged (18-70 years) of both sexes

Exclusion Criteria:

* History or current evidence of any CNS disease other than SAH which may cause cardiac complications.
* History or current evidence of medical illness as endocrinal and metabolic disorders which may cause cardiac complications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presented with spontaneous subarachnoid hemorrhage admitted to our department included in this study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Electrocadriogram | 1 miute
  to measure heart rate (beats/minute) in subarachnoid hemorrhage patients
Echocardiogarphy | 30 minute
  to measure ejection fraction (%) in subarachnoid hemorrhage patients

SECONDARY OUTCOMES:
serum treponin level | 30 minute
  to measure serum treponin(ng/ml)in subarachnoid hemorrhage patients